CLINICAL TRIAL: NCT04779905
Title: Assessment of Chronic Kidney Disease in Non Alcoholic Fatty Liver Disease(NAFLD) Patients
Brief Title: Chronic Kidney Disease and Non-alcoholic Fatty Liver Diseases
Acronym: NAFLD
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mona Mohammed Abdelrhman, Principal investigator, Sohag University
Other Study IDs: Soh-Med-21-02-40
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Chronic Kidney Diseases; NAFLD
Keywords: chronic kidney disease; NAFLD; Hepatic fibrosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-alcoholic Fatty Liver Diseases: patients diagnosed to has NAFLD by ultrasonography presented to the outpatient clinic of Sohag University Hospital
  Interventions: Diagnostic Test: urinary albumbin/creatinine ratio
- control: healthy volunteers who looks normal on ultrasonography
  Interventions: Diagnostic Test: urinary albumbin/creatinine ratio

INTERVENTIONS:
Diagnostic Test: urinary albumbin/creatinine ratio — detection of microalbuminuria in nafld patients
  Other Names: estimated glomerular filtration rate

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease worldwide. This disease reportedly affects up to 30% of the general population in Western countries, especially in patients with metabolic syndrome, obesity, and type II diabetes. NAFLD is considered to be an independent risk factor for cardiovascular disease and there is accumulating evidence to support a causative role in the development of chronic kidney disease (CKD). So, we aim first to assess the prevalence of chronic kidney disease in NAFLD patients, secondly to detect the association between hepatic fibrosis and CKD in NAFLD patients

DETAILED DESCRIPTION:
This study will be conducted on 100 patients 70 patients diagnosed to has NAFLD by ultrasonography presented to the outpatient clinic of Sohag University Hospital, and A control group of 30 healthy volunteers who looks normal on ultrasonography from February 2021 to July 2021.

Methods:

All included patients will be subjected to:

1. Detailed history, complete general and systemic examination .
2. BMI will be calculated as follow
3. Abdominal Ultrasonography.
4. Laboratory investigations:

   Fasting and post-prandial blood sugar Serum lipogram. Liver function tests. Serum creatinine, Albumin -creatinine Ratio.
5. Calculation of estimated Glomerular Filtration Rate eGFR.
6. Liver stiffness measurements to detect degree of fibrosis and measurement of the degree of steatosis using (Fibroscan)

Ethical considerations:

The study will be approved by The Ethical committee of Sohag Faculty of Medicine, Sohag University.

The study protocol will be adherent to practice guidelines of the World Medical Association Code of Ethics (Declaration of Helsinki).

After explanation about the nature of the procedures, possible complications, benefits, and steps of the study, All patients will give a written informed consent for participating in the study, performing abdominal ultrasound, taking blood samples, performing fibroscan.

ELIGIBILITY:
Inclusion Criteria:

patients diagnosed to has NAFLD by ultrasonography presented to the outpatient clinic of Sohag University Hospital

Exclusion Criteria:

1. Diabetic patients.
2. Hypertensive patients.
3. Other causes of chronic liver disease rather than NAFLD.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will be conducted on 100 patients 70 patients diagnosed to has NAFLD by ultrasonography presented to the outpatient clinic of Sohag University Hospital, and A control group of 30 healthy volunteers who looks normal on ultrasonography from February 2021 to July 2021
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
prevalence of chronic kidney disease in nafld patient | February 2021 to July 2021
correlation of chronic kidney disease and degree of hepatic fibrosis in nafld patient | February 2021 to July 2021

CONTACTS AND LOCATIONS:
Overall Officials: Radwa Farag, MD, Study Chair — Sohag University; Mohamed Amin, MD, Study Chair — Sohag University; Shimaa Hemdan, MD, Study Chair — Sohag University
Locations (1):
- Mona Mohammed Abdelrahman, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vernon G, Baranova A, Younossi ZM. Systematic review: the epidemiology and natural history of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis in adults. Aliment Pharmacol Ther. 2011 Aug;34(3):274-85. doi: 10.1111/j.1365-2036.2011.04724.x. Epub 2011 May 30. PMID 21623852
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-23. doi: 10.1002/hep.25762. No abstract available. PMID 22488764
- [Background] Loomba R, Sanyal AJ. The global NAFLD epidemic. Nat Rev Gastroenterol Hepatol. 2013 Nov;10(11):686-90. doi: 10.1038/nrgastro.2013.171. Epub 2013 Sep 17. PMID 24042449
- [Background] McCullough K, Sharma P, Ali T, Khan I, Smith WC, MacLeod A, Black C. Measuring the population burden of chronic kidney disease: a systematic literature review of the estimated prevalence of impaired kidney function. Nephrol Dial Transplant. 2012 May;27(5):1812-21. doi: 10.1093/ndt/gfr547. Epub 2011 Sep 29. PMID 21965592